CLINICAL TRIAL: NCT00782652
Title: The Effects of Nitric Oxide for Inhalation on Survival or the Need for Dialysis or a Right Ventricular Assistance Device (RVAD) in Right Ventricular Infarction Patients
Brief Title: The Effects of Nitric Oxide for Inhalation in Right Ventricular Infarction Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INOT43
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Right Ventricular Infarction
Keywords: myocaridal infarction; right ventricular infarction; cardiogenic shock; RVAD; Right ventricular assist device; cardiac disease; right ventricle; cardiac shock; heart dysfunction
MeSH Terms: conditions — Shock, Cardiogenic; Heart Diseases | interventions — Endothelium-Dependent Relaxing Factors; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): inhaled nitric oxide at 40 or 80ppm
  Interventions: Drug: inhaled nitric oxide
- 2 (Placebo Comparator): inhaled nitrogen at either 40 or 80ppm
  Interventions: Drug: nitrogen gas

INTERVENTIONS:
Drug: inhaled nitric oxide — Continuous delivery at either 40 or 80 ppm for a duration of up to 14 days
  Other Names: INOmax
  Arms: 1
Drug: nitrogen gas — Continuous delivery at either 40 or 80 ppm for a duration of up to 14 days
  Arms: 2

SUMMARY:
This study is designed to better understand the effects of nitric oxide, a gas for inhalation, on patients with right ventricular infarction.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, placebo-controlled study that will assess the feasibility of studying inhaled nitric oxide for the treatment of cardiogenic shock due to right ventricular infarction, and the dose response of the acute hemodynamic changes occurring with nitric oxide inhalation in these patients. Patients with evidence of right ventricular infarction and cardiogenic shock, and have angiographic evidence of impaired blood flow to the right ventricle, or if right ventricular coronary perfusion is unimpared, cardiac shock persists, will be eligible for enrollment. Patients will receive standard of care for their condition, and will also recieve either nitric oxide for inhalation or placebo for up to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Acute inferior mycardial infarction (defined as an episode of chest pain lasting >30 minutes and electrocardiographic evidence of 1 mm or greater ST elevation in inferior leads) within the past 72 hours.
* Invasive hemodynamic evidence of hemodynamically-significant RV dysfunction, defined as the presence of all the following: systemic venous congestion (mean RA pressure > 10mmHg), the ratio of RA/PCW pressure 0.75 or greater, a low cardiac output as determined by Fick or Thermodilution (TD) technique (cardiac index < 2.5 l/min/m2), systolic systemic arterial blood pressure of 90mmHg or less or requiring vasopressor or mechanical support to maintain systolic pressure > 90mmHg. Patients with a PCWP of 14mmHg or less should receive intravascular volume repletion until their PCWP is > 14mmHg.
* Coronary angiography revealing either an occlusion of the RCA proximal to any RV marginal branch or evidence of diminished flow to RV marginal branches of the RCA.
* If patient undergoes coronary revascularization, there must be evidence of unsuccessful right ventricular reperfusion (lack of restoration of TIMI grade III flow in the distal RCA and > 1mm RV marginal branches) or evidence of hemodynamically significant RVI must persist for greater than 1 hour after successful revascularization.
* Age 18 years or greater

Exclusion Criteria:

* PCW 25mmHg or greater or mechanical complications of myocardial infarction requiring surgical correction.
* Severe LV systolic dysfunction as determined by the principal investigator. Unprotected left main coronary stenosis > 50%.
* Pulmonary infiltrates consistent with pulonary edema on chest X-ray (if chest X-ray is clinically indicated).
* Evidence of shock-related end-organ damage, including creatinine 3.0 or greater, metabolic acidosis (pH 7.1 or less) and not corrected by 100 ml NaHCO3 (1mEq/ml), disseminated intravascular coagulation, or clinical evidence of diffuse brain injury.
* Previous history of severe pericardial, congenital, or valvular heart disease.
* Refractory hemodynamically significant arrhythmia.
* Presence of pneumonia, adult respiratory distress syndrome, or sepsis.
* Prior history of pulmonary disease requiring chronic oxygen therapy.
* Pregnancy
* Use of investigational drugs or device within the 30 days prior to enrollment to the study.
* Uncontrolled active bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-03; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
survival to hospital discharge or Day 30, whichever occurs first without the need for renal replacement therapy or a Right Ventricular Assistance Device (RVAD) | hospital discharge or Day 30

SECONDARY OUTCOMES:
survival at 1 year after initial hospitalization | 1 year post treatment
time on vasoconstrictor or inotropic medications | study duration
duration of intraaortic balloon pump support, if applicable | study duration
time in intensive care unit | study duration
duration or need for mechanical ventilation | study duration
change in cardiac index by dose | baseline, hour 8, days 3 & 7, and at day 30 or discharge
change in right ventricule function and size by dose | baseline, hour 8, days 3 & 7 and at day 30 or discharge
change in pulmonary vascular resistance by dose | study duration
change in any right-to-left intracardiac shunt flow, as assessed by contrast echocardiography | study duration
neurohormonal assessment of prognosis with BNP, NT-pro BNP | Baseline, hour 8 and days 3 & 7
incidence of mortality | treatment duration through 1 year
incidence and types of reported adverse events | study duration through day 30 or discharge

CONTACTS AND LOCATIONS:
Locations (6):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
- University Hospital Gasthuisberg, University of Leuven, Leuven, Belgium
- Univeristy of Ottawa Heart Institute, Ottawa, Ontario, Canada
- Institute of Cardiology Warsaw, Alpejska, Poland
- Cardiovascular Department, Hospital Clinic, Barcelona, Spain